CLINICAL TRIAL: NCT01952821
Title: The Validity and Reliability of the Six-Minute Walk Test, Ten-Meter Walk Test, 30 Second Chair Stand, Linear Analog Scale of Function, and the Modified Brief Fatigue Inventory in Patients With Cancer of the Head and Neck
Brief Title: Validity and Reliability of Outcome Measures in Patients With Cancer of the Head and Neck
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Melissa M. Eden, Physical Therapist, Mayo Clinic
Other Study IDs: 13-004891
Record Dates: First submitted 2013-09-21; First posted 2013-09-30 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Physical function; Cancer Related Fatigue; Gait Speed; 6MWT; 10-Meter Walk Test; 30-Second Chair Stand; Linear Analog Scale of Function; Modified Brief Fatigue Inventory
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Test Group: This group will receive all listed outcome measures on 2 testing visits.
  Interventions: Other: Six-Minute Walk Test; Other: 10-Meter Walk Test; Other: 30-Second Chair Stand; Other: Linear Analog Scale of Function; Other: Modified Brief Fatigue Inventory; Other: FACIT-Fatigue

INTERVENTIONS:
Other: Six-Minute Walk Test
Other: 10-Meter Walk Test
Other: 30-Second Chair Stand
Other: Linear Analog Scale of Function
Other: Modified Brief Fatigue Inventory
Other: FACIT-Fatigue

SUMMARY:
The purpose of this study is to establish the Six-Minute Walk Test, 10-Meter Walk Test, 30 Second Chair Stand, Linear Analog Scale of Function, and the Modifed Brief Fatigue Inventory as reliable and valid outcome measurements for patients with head and neck cancer.

DETAILED DESCRIPTION:
This study will be looking at the test-retest reliability and validity of various outcome measures in patients with cancer of the head and neck. Testing will occur in 2 visits within one week.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Within 3 months of surgery, or are currently undergoing radiation and/or chemotherapy for a diagnosis of head and neck cancer
* Community dwelling
* Able to provide informed consent, answer relevant questionnaires,follow instructions provided during testing

Exclusion Criteria:

* Vulnerable populations (minors, prisoners)
* Medical comorbidities which limit the safe completion of the 6MWT, gait speed, and strength testing
* Inability to return for a second day of testing within one week

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling patients with a new or recurrent diagnosis of head and neck cancer.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Six-Minute Walk Test | Baseline - 1 week
10-Meter Walk Test | Baseline - 1 week
30-Second Chair Stand | Baseline - 1 week
Linear Analog Scale of Function | Baseline - 1 week
Modified Brief Fatigue Inventory | Baseline - 1 week

SECONDARY OUTCOMES:
FACIT-Fatigue | Baseline - 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M. Eden, DPT, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States